CLINICAL TRIAL: NCT02785185
Title: A Phase 2, Multi-Center, Double-Blind, Randomized, Vehicle-Controlled Study to Compare the Safety and Efficacy of IDP-122 Lotion (0.01% Halobetasol Propionate) to Ultravate® (Halobetasol Propionate) Cream, in the Treatment of Plaque Psoriasis
Brief Title: Safety and Efficacy of IDP-122 Lotion When Applied Topically to Subjects With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V01-122A-203
Record Dates: First submitted 2016-04-26; First posted 2016-05-27 (Estimated); Results first posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — halobetasol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- IDP-122 Lotion (Experimental): Lotion
  Interventions: Drug: IDP-122 Lotion
- Ultravate Cream (Active Comparator): Cream
  Interventions: Drug: Ultravate Cream
- IDP-122 Vehicle Lotion (Active Comparator): Lotion
  Interventions: Drug: IDP-122 Vehicle Lotion
- IDP-122 Vehicle Cream (Active Comparator): Cream
  Interventions: Drug: IDP-122 Vehicle Cream

INTERVENTIONS:
Drug: IDP-122 Vehicle Lotion — Vehicle
  Other Names: Lotion
  Arms: IDP-122 Vehicle Lotion
Drug: IDP-122 Vehicle Cream — Vehicle
  Other Names: Cream
  Arms: IDP-122 Vehicle Cream
Drug: IDP-122 Lotion — Lotion
  Other Names: Lotion
  Arms: IDP-122 Lotion
Drug: Ultravate Cream — Cream
  Other Names: Ultravate
  Arms: Ultravate Cream

SUMMARY:
A Phase 2, Multi-Center, Double-Blind, Randomized, Vehicle-Controlled Study.

DETAILED DESCRIPTION:
A Phase 2, Multi-Center, Double-Blind, Randomized, Vehicle-Controlled Study to Compare the Safety and Efficacy of IDP-122 Lotion (0.01% halobetasol propionate) to Ultravate® (halobetasol propionate) Cream, 0.05% in the Treatment of Plaque Psoriasis.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female, of any race, at least 18 years of age (inclusive).
* Freely provides both verbal and written informed consent.
* Is willing and able to avoid prolonged exposure of the treatment area to ultraviolet radiation (natural and artificial) for the duration of the study.
* Subject is willing to comply with study instructions and return to the clinic for required visits.

Key Exclusion Criteria:

* Has spontaneously improving or rapidly deteriorating plaque psoriasis or pustular psoriasis, as determined by the investigator.
* Presents with psoriasis that was treated with prescription medication and failed to respond to treatment, even partially or temporarily, as determined by the investigator.
* Presents with any concurrent skin condition that could interfere with the evaluation of the treatment areas, as determined by the investigator.
* Is pregnant, nursing an infant, or planning a pregnancy during the study period.
* Has received treatment with any investigational drug or device within 60 days or 5 drug half-lives (whichever is longer) prior to the Baseline visit, or is concurrently participating in another clinical study with an investigational drug or device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-12-02 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Binu J Alexander, MD, Study Director — Valeant Pharmaceuticals
Locations (13):
- United States (13):
  - Valeant Site 05, Rogers, Arkansas
  - Valeant Site 10, Beverly Hills, California
  - Valeant Site 09, Carlsbad, California
  - Valeant Site 13, Los Angeles, California
  - Valeant Site 12, Santa Monica, California
  - Valeant Site 07, Coral Gables, Florida
  - Valeant Site 11, North Miami Beach, Florida
  - Valeant Site 03, Sanford, Florida
  - Valeant Site 08, Albany, Indiana
  - Valeant Site 04, Louisville, Kentucky
  - Valeant Site 06, Fridley, Minnesota
  - Valeant Site 02, High Point, North Carolina
  - Valeant Site 01, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Kerdel FA, Draelos ZD, Tyring SK, Lin T, Pillai R. A phase 2, multicenter, double-blind, randomized, vehicle-controlled clinical study to compare the safety and efficacy of a halobetasol propionate 0.01% lotion and halobetasol propionate 0.05% cream in the treatment of plaque psoriasis. J Dermatolog Treat. 2019 Jun;30(4):333-339. doi: 10.1080/09546634.2018.1523362. Epub 2018 Nov 5. PMID 30207807

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IDP-122 Lotion | Ultravate Cream | IDP-122 Vehicle Lotion | IDP-122 Vehicle Cream
Started | 60 | 57 | 17 | 16
Completed | 59 | 56 | 15 | 16
Not Completed | 1 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDP-122 Lotion | Ultravate Cream | IDP-122 Vehicle Lotion | IDP-122 Vehicle Cream | Total
Number analyzed (Participants) | 60 | 57 | 17 | 16 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (14.2) | 50.2 (10.91) | 44.7 (8.8) | 48.6 (14.98) | 49.6 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 27 | 6 | 12 | 70
  Male | 35 | 30 | 11 | 4 | 80

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Success of a 2-Grade IGA Score Improvement From Baseline and an IGA Score of Clear or Almost Clear at Week 2
Description: Treatment success defined as at least a 2-grade improvement from Baseline in the Investigator's Global Assessment (IGA) score and an IGA score equating to "clear" or "almost clear" at Week 2. The IGA score was based on a 5-point scale ranging from 0 to 4 (0=clear, 1=almost clear, 2=mild, 3=moderate, and 4=severe).
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | IDP-122 Lotion | Ultravate Cream | IDP-122 Vehicle Lotion | IDP-122 Vehicle Cream
Number analyzed (Participants) | 60 | 57 | 17 | 16
Participants | 18 | 18 | 3 | 1

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Adverse events were collected from participants who were randomized, received at least 1 confirmed dose of study drug, and had at least 1 post-Baseline safety assessment (Safety Population).
Arm/Group | IDP-122 Lotion | Ultravate Cream | IDP-122 Vehicle Lotion | IDP-122 Vehicle Cream
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/57 | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 0/60 | 0/57 | 1/15 | 0/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IDP-122 Lotion (N=60) | Ultravate Cream (N=57) | IDP-122 Vehicle Lotion (N=15) | IDP-122 Vehicle Cream (N=16)
Application site warmth (General disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.